CLINICAL TRIAL: NCT06504615
Title: A French, Prospective, Observational, Multicenter Study of Patients Treated With Nivolumab Plus Chemotherapy as First Line Treatment in Advanced or Metastatic Esophageal Squamous Cell Carcinoma, Esophageal Adenocarcinoma, Gastroesophageal Junction Adenocarcinoma or Gastric Adenocarcinoma [METAGIO]
Brief Title: Observational Study of Patients Treated With Nivolumab and Chemotherapy for Advanced or Metastatic Esophageal, Gastroesophageal or Gastric Cancer in France
Acronym: METAGIO
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-1408
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Gastric Adenocarcinoma; Gastro-esophageal Junction Adenocarcinoma; Esophageal Adenocarcinoma (EAC); Esophageal Squamous Cell Carcinoma (ESCC)
Keywords: Gastric adenocarcinoma; Gastro-esophageal junction (GEJ) adenocarcinoma; Esophageal adenocarcinoma (EAC); Esophageal squamous cell carcinoma (ESCC)
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma; Adenocarcinoma | interventions — Nivolumab; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Participants with a diagnosis of gastric adenocarcinoma, gastro-esophageal junction adenocarcinoma or esophageal adenocarcinoma
  Interventions: Drug: nivolumab + chemotherapy
- Cohort 2: Participants with a diagnosis of untreated, unresectable, advanced, recurrent, or metastatic esophageal squamous cell carcinoma
  Interventions: Drug: nivolumab + chemotherapy

INTERVENTIONS:
Drug: nivolumab + chemotherapy — As prescribed by the treating clinician, as per product label

SUMMARY:
A study to estimate the overall survival in real-life conditions in France of adult participants treated with nivolumab in combination with chemotherapy as first-line treatment for gastric and gastroesophageal junction cancer.

ELIGIBILITY:
Inclusion Criteria:

Cohorts 1 & 2

* Adult participants (at least 18 years of age at time of treatment decision)
* Participants treated with nivolumab in combination with fluoropyrimidine- and platinum-based chemotherapy (according to the French current marketing authorization) for the treatment of Gastric Adenocarcinoma, Gastro-Esophageal Junction (GEJ) adenocarcinoma, Esophageal Adenocarcinoma (EAC) or Esophageal Squamous Cell Carcinoma (ESCC) and prior to study participation.
* Participants who provided oral informed consent to participate in the study

Cohort 1 only • Diagnosis of untreated HER2 negative advanced or metastatic gastric adenocarcinoma, GEJ adenocarcinoma or EAC whose tumor express PD-L1 with a CPS ≥5

Cohort 2 only

• Diagnosis of untreated unresectable advanced, recurrent or metastatic ESCC with tumor cell PD-L1 expression (TPS) ≥1%

Exclusion Criteria:

Cohorts 1 & 2

* Participants with a primary diagnosis of a cancer other than advanced or metastatic gastric adenocarcinoma, GEJ adenocarcinoma, EAC or ESCC, within the past 5 years.
* Participants currently enrolled in an interventional clinical trial for his/her advanced or metastatic gastric adenocarcinoma, GEJ adenocarcinoma, EAC or ESCC.
* Pregnant women
* Participants under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants in France diagnosed with Gastric Adenocarcinoma, Gastro-Esophageal Junction (GEJ) adenocarcinoma, Esophageal Adenocarcinoma (EAC) or Esophageal Squamous Cell Carcinoma (ESCC) and treated with nivolumab in combination with fluoropyrimidine- and platinum-based chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Day 0 and months 2-3, 4-6, 8-9, 12, 18, 24, 30 and 36

SECONDARY OUTCOMES:
Cause of death (where available) | Day 0 and months 2-3, 4-6, 8-9, 12, 18, 24, 30 and 36
Disease progression | Day 0 and months 2-3, 4-6, 8-9, 12, 18, 24, 30 and 36
  As assessed by the Site Investigator
Progression-free survival (PFS) | Day 0 and months 2, 3, 4-6, 8-9, 12, 18, 24, 30 and 36
Time to treatment discontinuation (TTD) | Day 0 and months 2-3, 4-6, 8-9, 12, 18, 24, 30 and 36
Time to failure of strategy (TFS) | Day 0 and months 2-3, 4-6, 8-9, 12, 18, 24, 30 and 36
Time to next Treatment (TTNT) | Day 0 and months 2-3, 4-6, 8-9, 12, 18, 24, 30 and 36
Second progression-free survival (PFS2) | Day 0 and months 2-3, 4-6, 8-9, 12, 18, 24, 30 and 36
Treatment Free Interval (TFI) | Day 0 and months 2-3, 4-6, 8-9, 12, 18, 24, 30 and 36
Overall tumor response (ORR) | Day 0 and months 2-3, 4-6, 8-9, 12, 18, 24, 30 and 36
Response rate | Day 0 and months 2-3, 4-6, 8-9, 12, 18, 24, 30 and 36
Duration of response (DOR) | Day 0 and months 2-3, 4-6, 8-9, 12, 18, 24, 30 and 36
Participant socio-demographics | Baseline
Participant clinical characteristics | Baseline
Participant treatment history | Baseline
Nivolumab treatment regime | Day 0 and months 2-3, 4-6, 8-9, 12, 18, 24, 30 and 36
Chemotherapy treatment regime | Day 0 and months 2-3, 4-6, 8-9, 12, 18, 24, 30 and 36
Reason for treatment discontinuation | Day 0 and months 2-3, 4-6, 8-9, 12, 18, 24, 30 and 36
Subsequent non-systemic treatment received post first-line treatment | Day 0 and months 2-3, 4-6, 8-9, 12, 18, 24, 30 and 36
Subsequent systemic treatment received post first-line treatment | Day 0 and months 2-3, 4-6, 8-9, 12, 18, 24, 30 and 36
Subsequent systemic treatment effectiveness | Day 0 and months 2-3, 4-6, 8-9, 12, 18, 24, 30 and 36
Participant adverse events (AEs) | Up to 3 years
Participant health related quality of life as assessed by 5-level EuroQoL-5 dimension version (EQ-5D-5L) | Day 0 and months 2-3, 4-6, 8-9, 12, 18, 24, 30 and 36

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- France (2):
  - KAPPA SANTE Institution, Paris
  - Kappa Santé, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts